CLINICAL TRIAL: NCT06318208
Title: Pulmonary Function in Non-hospitalized Adults and Children After Mild COVID-19
Status: Completed | Type: Observational
Sponsor: University of Rostock (Other)
Responsible Party: Principal Investigator, Alexandra Rachel Görges, Principal Investigator, University of Rostock
Other Study IDs: C-LCI
Record Dates: First submitted 2024-03-17; First posted 2024-03-19 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: SARS-CoV-2 Infection
Keywords: mild COVID-19; LCI; lung function; non-hospitalized COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: lung function testing — lung function testing including LCI, FEV1, FVC, DLCO

SUMMARY:
The study investigates whether patients with mild SARS-CoV-2 infection, who stayed at home during their infection and weren't hospitalized, have any persisting sequelae in pulmonary function.

Therefore, 110 patients, aged 6-60 years, were recruited by telephone 4-12 weeks after laboratory-confirmed positive PCR and invited for a lung function testing. Every patient with abnormalities in pulmonary function was invited to a follow-up 3 months after the first appointment to assess changes in lung function values.

Patients with a pre-existing lung disease and smokers within the last five years were excluded beforehand.

Additionally to lung function testing we did a throat swab at each appointment to analyse via Multiplex PCR whether the patients had any other respiratory infection at the time of the pulmonary function testing.

DETAILED DESCRIPTION:
110 patients, 90 adults and 20 children, were recruited. The lung function included LCI, FEV1, FVC and DLCO (Hb corrected). Additionally we did a throat swab at each appointment to analyse via Multiplex PCR whether the patients had any other respiratory infection at the time of the test.

ELIGIBILITY:
Inclusion Criteria:

* SARS-CoV-2 Infection, non-hospitalized during infection

Exclusion Criteria:

* Smoking, existing lung disease (COPD, Asthma bronchiale)

Ages: 6 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: SARS-Covid -2 Infection 1 months before investigation
Sampling Method: Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2021-04-20 (Actual); Primary Completion 2022-01-03 (Actual); Study Completion 2022-01-03 (Actual)

PRIMARY OUTCOMES:
Pulmonary function | 4.3 - 11.3 weeks after positive PCR for SARS-CoV-2
  Pulmonary function after SARS-CoV-2 Infection

SECONDARY OUTCOMES:
Changes in pulmonary function | 11.0 - 16.7 weeks after the first lung function testing
  Changes in pulmonary function towards the follow-up
Sociodemographic factors | 9 months
  Relation of pulmonary function to sociodemographic factors

CONTACTS AND LOCATIONS:
Overall Officials: Manfred Ballmann, Prof. Dr., Study Director — UMR Kinder- und Jugendklinik
Locations (1):
- Kinder- und Jugendklinik Universitätsmedizin Rostock, Rostock, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gorges AR, Warnke P, Lobermann M, Zapf A, Weitzel J, Steinbach ML, Zufle-Lemke N, Fischer DC, Ballmann M. Pulmonary function in non-hospitalized adults and children after mild COVID-19: a single-centre prospective cohort study. BMC Pulm Med. 2025 Nov 6;25(1):511. doi: 10.1186/s12890-025-04007-y. PMID 41199209